CLINICAL TRIAL: NCT01734226
Title: Efficacy and Safety of Prunus Mume Extract on Improvement of Constipation
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chonbuk National University Hospital (Other)
Responsible Party: Principal Investigator, Soo-Wan Chae, Principal Investigator, Clinical Trial Center for Functional Foods, Chonbuk National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: JINR-CON-PME
Record Dates: First submitted 2012-11-22; First posted 2012-11-27 (Estimated); Last update posted 2012-11-28 (Estimated); Status verified 2012-11

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Prunus Mume Extract (Experimental)
  Interventions: Dietary Supplement: Prunus Mume Extract
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Prunus Mume Extract — Prunus Mume Extract (3.94g/day)
  Arms: Prunus Mume Extract
Dietary Supplement: Placebo — Placebo (3.94g/day)
  Arms: Placebo

SUMMARY:
The investigators performed a 8-week, randomized, double-blind, placebo-controlled human trial to evaluate the efficacy and safety of Prunus Mume Extract on Improvement of Constipation. The investigators measured Improvement of Constipation parameters , including Colonic Transit Time, number of bowel movement, defecation time, stool type, color and stool amounts per defecation, and monitored their blood pressure.

ELIGIBILITY:
Inclusion Criteria:

* Males and females 19-40 years old
* Subject who have functional constipation by ROME IIII criteria
* Subject who have over 36 hour colonic transit time
* Able to give informed consent

Exclusion Criteria:

* Subject who have Irritable bowel syndrome by ROME IIII criteria
* Allergic or hypersensitive to any of the ingredients in the test products
* History of reaction to any of the test products or of gastrointestinal diseases such as Crohn's disease or gastrointestinal surgery
* History of alcohol or substance abuse
* Participation in any other clinical trials within past 2 months
* Laboratory test, medical or psychological conditions deemed by the investigators to interfere with successful participation in the study
* Pregnant or lactating women etc.

Ages: 19 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2012-08; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Estimated)

PRIMARY OUTCOMES:
Changes in Colonic Transit Time | 8 weeks
  Colonic Transit Time was measured in study visit 1(0 week) and visit 3(8 week).
Changes in number of bowel movement | 8 weeks
  Number of bowel movement was measured in study visit 1(0 week) and visit 3(8 week).
Changes in defecation time | 8 weeks
  Defecation time was measured in study visit 1(0 week) and visit 3(8 week).

SECONDARY OUTCOMES:
Changes in stool type | 8 weeks
  Stool type was measured in study visit 1(0 week) and visit 3(8 week).
Changes in stool color | 8 weeks
  Stool color was measured in study visit 1(0 week) and visit 3(8 week).
Changes in stool amounts per defecation | 8 weeks
  Stool amounts per defecation was measured in study visit 1(0 week) and visit 3(8 week).

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical Trial Center for Functional Foods; Chonbuk National University Hospital, Jeonju, Jeollabuk-do, South Korea